CLINICAL TRIAL: NCT06657612
Title: Is Ultrasound-Guided Steroid Injection Less Effective in Carpal Tunnel Syndrome Patients with Bifid Median Nerve?: a Focus on Short-Term Efficacy
Brief Title: Is Ultrasound-Guided Steroid Injection Less Effective in Carpal Tunnel Syndrome Patients with Bifid Median Nerve?
Status: Completed | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH6
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bifid median nerve: Patients (diagnosed with carpal tunnel syndrome) with bifid median nerve
  Interventions: Other: No intervention
- Control group: Patients (diagnosed with carpal tunnel syndrome) with normal median nerve
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study is to evaluate the short-term efficacy of ultrasound-guided corticosteroid injection in patients with and without bifid median nerve.

DETAILED DESCRIPTION:
Twenty-five patients with bifid median nerve and twenty-five patients without bifid median nerve, aged 18-65, who applied to the Physical Therapy and Rehabilitation outpatient clinic at Beylikdüzü State Hospital, diagnosed with mild to moderate carpal tunnel syndrome based on electrophysiological studies, and who received ultrasound-guided corticosteroid injection, will be included in our study. Patients identified as having a bifid median nerve during the injection will be noted and invited for a follow-up at the 1st month to assess their pain and functional status. The same follow-up visit will be conducted for an equal number of age- and gender-matched patients without bifid median nerve who received the injection. At the end of the study, the 1-month efficacy of the injection in both groups will be evaluated. Patients who agree to participate in the study will be asked to complete the Visual Analog Scale (VAS), the Boston Carpal Tunnel Syndrome Questionnaire (BCTQ), and the Quick Disabilities of the Arm, Shoulder, and Hand Questionnaire (Quick-DASH) before the injection. They will then be invited for a follow-up visit at the 1st month, where the VAS, BCTQ, and Quick-DASH will be administered again.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65.
* Diagnosed with mild to moderate carpal tunnel syndrome based on electrophysiological studies conducted within the last 6 months.
* Scheduled for ultrasound-guided corticosteroid injection.
* Patients who have agreed to participate in the study.

Exclusion Criteria:

* Diagnosis of any other condition that could cause neuropathic symptoms, such as polyneuropathy, brachial plexopathy, or thoracic outlet syndrome.
* Previous history of injection or surgery for carpal tunnel syndrome
* Patients who refuse to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild to moderate carpal tunnel syndrome
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS): | 0 day, 4th week
  The Visual Analog Scale is a widely used tool to assess the intensity of pain. It consists of a straight line, typically 10 cm in length, where one end represents "no pain" (0) and the other end represents "worst imaginable pain" (10). Patients mark a point on the line that corresponds to their current level of pain. VAS provides a simple, quantitative measure of pain that is easy for patients to use and for clinicians to interpret, making it a reliable tool for tracking changes in pain levels over time.
Boston Carpal Tunnel Syndrome Questionnaire Symptom Severity Scale (BCTQ-SSS): | 0 day, 4th week
  The SSS assesses the severity of carpal tunnel symptoms such as pain, tingling, and numbness. The total score for this scale ranges from a minimum of 11 to a maximum of 55. A lower score indicates mild or no symptoms, while a higher score suggests more severe symptoms. As the score increases, the severity of symptoms worsens, with a score closer to 55 reflecting a significantly greater impact on daily life.
Quick Disabilities of the Arm, Shoulder, and Hand Questionnaire (Quick-DASH): | 0 day, 4th week
  The Quick-DASH is a shortened version of the full DASH questionnaire, designed to measure physical function and symptoms in people with musculoskeletal disorders of the upper limb. It consists of 11 items that assess the difficulty a patient experiences in performing activities of daily living, such as carrying a heavy object, opening a jar, or using a computer. Each item is scored on a 5-point Likert scale, where higher scores reflect greater disability. The Quick-DASH is a validated, efficient tool that provides a broad overview of the patient's upper extremity function and how their condition affects daily life.
Boston Carpal Tunnel Syndrome Questionnaire Functional Status Scale (BCTQ-FSS): | 0 day, 4th week
  The FSS evaluates how carpal tunnel syndrome affects a person's ability to perform daily tasks like writing, buttoning clothes, or holding objects. The total score for this scale ranges from a minimum of 8 to a maximum of 40. A lower score suggests little to no difficulty in performing these tasks, while a higher score reflects greater functional limitations. As the FSS score increases, it indicates that the condition is having a more pronounced effect on daily functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No